CLINICAL TRIAL: NCT06240676
Title: Examining the Effect of Breastfeeding Education Given to Mothers Based on Postpartum Awareness Practices on Breast Milk and Cortisol Hormone at the Newborn Circadian Level
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kafkas University (Other)
Responsible Party: Principal Investigator, Şevin Akgün, research assistant, Kafkas University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KAU-HEM-SA-01
Record Dates: First submitted 2024-01-17; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Mother Fetus Relations; Health Behavior
Keywords: Breast Milk, Cortisol Hormone, Conscious Awareness, Stress
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Intervention Model Description: THE FEMALE MILK OF TWO GROUPS WILL BE COMPARED WITH EDUCATIONAL AND NON-EDUCATIONAL
Who Masked: Participant
Masking Description: Participants will be given the option of two envelopes, one of which is experiment and the other is control. Participants will be asked to choose one of the two envelopes when applying to the obstetrics clinic of the hospital.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): After the 3rd month postpartum, mothers who are given classical breastfeeding training by the researcher will then be given a breastfeeding training based on mindfulness therapy methods. After the classical breastfeeding training, a pre-test will be applied and then mindfulness-based training will be started. The effectiveness of the training will also be determined within the group with the post-test to be applied after the training. A sleep diary will be applied to the newborn. After breastfeeding, how many hours of sleep and body temperature will be noted.
  Interventions: Behavioral: AWARENESS-BASED COGNITIVE THERAPY
- control group (No Intervention): From mothers whose information was collected during pregnancy, only breast milk will be taken for 1 week without any intervention in the 3rd month after birth.

INTERVENTIONS:
Behavioral: AWARENESS-BASED COGNITIVE THERAPY — A 6-week training program based on mindfulness practices will be applied to the experimental group determined by the single-blind method, after the 3rd month after birth. In order to observe the change in the experimental group, breast milk will be taken for pre-test (morning and evening) before training. After 6 weeks of training, a cortisol test will be performed by taking breast milk at 09:00 in the morning and 09:00 in the evening. Taken milk will be stored in the deep freezer for 1 week at -18 degrees. After the samples are prepared for testing under appropriate conditions (centrifuge), biochemical measurements will be made and recorded with the help of the SUNREDBIO brand human cortisol kit (the serial number is not known since we did not purchase the cortisol kit).A sleep diary will be used to measure newborn circadian rhythm.
  Arms: experimental group

SUMMARY:
In addition to being an easily accessible and ready-made food for babies in the first years of life, breast milk plays a major role in transmitting information about the time of day to newborn babies and therefore in the formation of the circadian rhythm, thanks to the hormones and various immune elements it contains.The main theme of mindfulness-based programs is mind and body meditation by focusing on the present moment, directing perception to inner experiences and observing these experiences.Regular practice of this type of meditation contributes greatly to increasing happiness and developing positive attitudes such as insight, compassion, awareness and stress management.Cortisol is the main stress hormone in the human body and is therefore a promising benchmark for investigating the effects of mindfulness programs. The purpose of mindfulness-based breastfeeding training to be given to mothers; It is to contribute to a healthy and safe postpartum period and breastfeeding experience for the mother and the newborn by minimizing the negative effects of the postpartum stress level in the mother and the cortisol hormone levels transferred from the mother's milk to the baby on the circadian rhythm.For this purpose, the sample size was planned to be a total of 54 people, 27 people per group, in the experimental design, with G power 3.1 analysis. The research will be conducted on healthy breastfeeding mothers who applied to Erzurum City Hospital and Kars Selim District State Hospital between 15.05.2023 and 15.06.2024.Subjects to be included in the study will be randomly selected among the pregnant women who applied to the clinic according to meeting the inclusion criteria. Breastfeeding: 'The Key to Sustainable Development'. For this reason, it is planned that the determination of the relationship between breast milk and circadian rhythm can be supported by cognitive methods, it will be important in terms of promoting breastfeeding and achieving development goals in a short time, and it is planned to contribute to the literature.

DETAILED DESCRIPTION:
In addition to being an easily accessible and ready-made food for babies in the first years of life, breast milk plays a major role in the transmission of information about the time of day to newborn babies, and therefore in the formation of circadian rhythm, thanks to the hormones and various immune elements it contains . Breast milk is the best way to convey information such as what time of day it is, when to go to sleep and when to wake up . Apart from this, transferring this information to the newborn in a unique way and ensuring its continuity is not as effective and easy as breast milk. The fact that the melatonin hormone, which rises in the breast milk in the evening hours, stimulates the smooth muscles and creates a resting effect, the increase in activity and the awakening state due to the effect of the cortisol hormone in the breast milk in the first hours of the day, ensures the formation of a regular sleep rhythm in the newborn.

Circadian rhythm regulates various physiological and psychological events in living organisms, such as sleep/wake rhythms, body temperature, blood pressure, hormone (melatonin, cortisol, etc.) synthesis and release, in a total period of 24 hours . Circadian rhythm continues to develop in the first three months of life. It is essential for the temporal adaptation process of the newborn and especially for mother-infant coordination . Delay or disruption of this situation negatively affects the neurocognitive development of the baby and causes metabolic problems as well as sleep problems . The most commonly used biological phase markers to examine circadian rhythm; cortisol and melatonin, whose oscillations are quite rhythmic . Cortisol acts through glucocorticoid receptors in almost all mammalian cells, helping to regulate the genetic clock in cells.Cortisol and melatonin levels in breast milk show parallelism with the levels of these hormones in the mother's plasma . The increase in cortisol levels in the first hours of the day and the increase in their rates in breast milk may affect the circadian rhythm negatively, instead of decreasing it in the following hours as a result of the continuity of the stress situation in the mother .

The main theme of mindfulness-based programs is mind and body meditation, which is formed by focusing on the present moment, directing the perception to inner experiences and observing these experiences . Regular practice of this type of meditation greatly contributes to increasing happiness and the development of positive attitudes such as insight, compassion, awareness, and stress management . Cortisol is the main stress hormone in the human body and is therefore a promising benchmark for investigating the effects of Mindfulness-Based Stress Reduction programs . In conjunction with other biological measures, the use of cortisol levels as a physiological marker of stress may be useful to confirm the self-reported benefits attributed to this program .

Among the recent studies on breast milk content on mothers and babies, cognitive-based approaches are preferred because they do not require intervention and have a low probability of posing a risk for the mother and baby, because they are easily accessible, and it is planned to obtain results that will contribute to the literature.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-35
* Having given birth at term (C/S and vaginal)
* Having a baby who is exclusively breastfed
* Not participating in any previous cognitive-based program
* Being at least literate
* No communication problems

Exclusion Criteria:

* Mothers with babies who have started supplementary feeding
* Having any health problems in mother and baby
* Premature baby
* Having given birth prematurely
* Illiteracy

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — mothers and expectant mothers
Enrollment: 54 (Estimated)
Dates: Start 2024-04-15 (Estimated); Primary Completion 2024-06-20 (Estimated); Study Completion 2024-06-20 (Estimated)

PRIMARY OUTCOMES:
measuring breast milk cortisol value | 4 MONTHS
  After 6 weeks of mindfulness-based breastfeeding training, the morning and evening values of the cortisol hormone in breast milk will be measured and compared with the breast milk of the group that was not trained.

SECONDARY OUTCOMES:
circadian rhythm of the newborn | 4 MONTHS
  Post-breastfeeding circadian rhythms (sleep-wakefulness) of babies of trained mothers will be evaluated through a sleep diary.

CONTACTS AND LOCATIONS:
Overall Officials: Rukiye TÜRK DELİBALTA, Study Director — Kafkas University Faculty Of Health Sciences; Şevin POLAT, Principal Investigator — Kafkas University Faculty Of Health Sciences
Locations (1):
- Kafkas Universty, Kars, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
For my study titled 'Investigation of the Effects of Breastfeeding Education Given to Mothers Based on Postpartum Mindfulness Practices on the Cortisol Hormone in Breast Milk and Newborn Circadian Levels', a signed document is obtained from the voluntary participants who participate in the study, stating that any information to be used in this study will not be shared with a third party.

REFERENCES:
- [Result] Creswell JD. Mindfulness Interventions. Annu Rev Psychol. 2017 Jan 3;68:491-516. doi: 10.1146/annurev-psych-042716-051139. Epub 2016 Sep 28. PMID 27687118
- [Result] Zollars I, Poirier TI, Pailden J. Effects of mindfulness meditation on mindfulness, mental well-being, and perceived stress. Curr Pharm Teach Learn. 2019 Oct;11(10):1022-1028. doi: 10.1016/j.cptl.2019.06.005. Epub 2019 Aug 7. PMID 31685171
- [Result] Parsons CE, Crane C, Parsons LJ, Fjorback LO, Kuyken W. Home practice in Mindfulness-Based Cognitive Therapy and Mindfulness-Based Stress Reduction: A systematic review and meta-analysis of participants' mindfulness practice and its association with outcomes. Behav Res Ther. 2017 Aug;95:29-41. doi: 10.1016/j.brat.2017.05.004. Epub 2017 May 10. PMID 28527330
- [Result] Ziomkiewicz A, Babiszewska M, Apanasewicz A, Piosek M, Wychowaniec P, Cierniak A, Barbarska O, Szoltysik M, Danel D, Wichary S. Psychosocial stress and cortisol stress reactivity predict breast milk composition. Sci Rep. 2021 Jun 2;11(1):11576. doi: 10.1038/s41598-021-90980-3. PMID 34078999
- [Result] Italianer MF, Naninck EFG, Roelants JA, van der Horst GTJ, Reiss IKM, Goudoever JBV, Joosten KFM, Chaves I, Vermeulen MJ. Circadian Variation in Human Milk Composition, a Systematic Review. Nutrients. 2020 Aug 4;12(8):2328. doi: 10.3390/nu12082328. PMID 32759654
- [Result] van der Voorn B, de Waard M, van Goudoever JB, Rotteveel J, Heijboer AC, Finken MJ. Breast-Milk Cortisol and Cortisone Concentrations Follow the Diurnal Rhythm of Maternal Hypothalamus-Pituitary-Adrenal Axis Activity. J Nutr. 2016 Nov;146(11):2174-2179. doi: 10.3945/jn.116.236349. Epub 2016 Sep 14. PMID 27629575
- [Result] Nagel EM, Howland MA, Pando C, Stang J, Mason SM, Fields DA, Demerath EW. Maternal Psychological Distress and Lactation and Breastfeeding Outcomes: a Narrative Review. Clin Ther. 2022 Feb;44(2):215-227. doi: 10.1016/j.clinthera.2021.11.007. Epub 2021 Dec 20. PMID 34937662